CLINICAL TRIAL: NCT02853058
Title: Uterine Artery Pulsatility Index During Labor After 34 Weeks in the Prediction of Materno Fetal Outcomes
Brief Title: Uterine Artery Pulsatility Index and Materno Fetal Outcomes
Acronym: UADLAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Amira Ayachi, University Assistant in Obstetrics and gynecology, University Tunis El Manar
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UTARTDOP1
Record Dates: First submitted 2016-07-24; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Labor Complication
Keywords: stillbirth; hemorrhage
MeSH Terms: conditions — Obstetric Labor Complications; Stillbirth; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal PI (Active Comparator): Uterine artery PI expresserd in MoM is <95e percentile
  Interventions: Radiation: normal PI
- pathological PI (Active Comparator): Uterine artery PI expressed in Multiple of Mediane (MoM) is >=95e percentile
  Interventions: Radiation: pathological PI

INTERVENTIONS:
Radiation: normal PI — measurement of the PI in the uterine artery for pregnant women during labor, expressed in MoM
  Arms: normal PI
Radiation: pathological PI — measurement of the PI in the uterine artery for pregnant women during labor, expressed in MoM
  Arms: pathological PI

SUMMARY:
High Uterine artery index pulsatility (PI) is associated with small for gestationnal age but also with stillbirth and distress during labor.

DETAILED DESCRIPTION:
measures of Uterine artery PI is made with transabdominal color flow during labor. The right and left uterine arteries are visualized at the crossover wth the external iliac arteries. PI is measured and the mean PI of the two vessels is calculated and expressed as multiple of the median (MoM).The outcomes stillbirth, distress and vaginal or cesarean delivery, apgar sore <7 at 5 minutes, birth weight and maternal outcomes: preeclampsia, hemorrhage and other complications are noted.

ELIGIBILITY:
Inclusion Criteria:

* gestationnal age >=34 weeks
* during labor

Exclusion Criteria:

* elective cesarean even if labor
* non elligible ultrasound criteria of good measurement of uterine artery PI

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
right uterine artery pulsatility index measurement | 15 minutes
left uterine artery pulsatility index measurement | 15 minutes

SECONDARY OUTCOMES:
maternal outcome | 2 days
  number of patients with hemorrhage, preeclampsie, adversal outcomes
small for gestationnal age (SGA) | 1 day
  number of neonatal SGA
Apgar Score<7 | 1 day
  number of birth with Apgar score <7
distress | 1 day
  number of cesarean section for distress

CONTACTS AND LOCATIONS:
Overall Officials: AMIRA AYACHI, Ph D, Study Chair — University Tunis El Manar
Locations (1):
- University Hospital Bougatfa, Bizerte, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valino N, Giunta G, Gallo DM, Akolekar R, Nicolaides KH. Uterine artery pulsatility index at 30-34 weeks' gestation in the prediction of adverse perinatal outcome. Ultrasound Obstet Gynecol. 2016 Mar;47(3):308-15. doi: 10.1002/uog.14898. Epub 2016 Feb 1. PMID 25970847